CLINICAL TRIAL: NCT06027593
Title: Using Electronically Derived AutoMated RePOrts of Appropriate Antibiotic Use to Inform SteWardship IntERventions
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-019749; 75D30121F00002 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 850722 (Other: University of Pennsylvania Institutional Review Board); 851400 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2023-08-14; First posted 2023-09-07 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Community-acquired Pneumonia; Acute Otitis Media; Pharyngitis
Keywords: Antibiotic stewardship; Implementation Science; Antibiotic Use; Outpatient antibiotic prescribing; Inpatient antibiotic prescribing
MeSH Terms: conditions — Community-Acquired Pneumonia; Otitis Media; Pharyngitis

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study measuring the impact of an antibiotic stewardship intervention consisting of clinician education and audit and feedback reports on antibiotic use for adult inpatients with community acquired pneumonia, pediatric inpatients with community acquired pneumonia, adult outpatients with acute pharyngitis, and pediatric outpatients with acute otitis media.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention: Patients diagnosed with conditions of interest during study period (No Intervention): Four population groups were included in the pre-intervention data: 1) adult inpatients with community acquired pneumonia; 2) pediatric inpatients with community acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media
- Post-Intervention: Patients diagnosed with conditions of interest during study period (Other): Four population groups were included in the post-intervention data: 1) adult inpatients with community acquired pneumonia; 2) pediatric inpatients with community acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media
  Interventions: Other: Quasi experimental intervention

INTERVENTIONS:
Other: Quasi experimental intervention — The intervention included clinician education and sharing of audit and feedback reports summarizing antibiotic use metrics for each of the four target conditions with treating clinicians.
  Arms: Post-Intervention: Patients diagnosed with conditions of interest during study period

SUMMARY:
The main goal of this study is to use automated electronic reports to assess and improve guideline-concordant antibiotic use for:

1) adult inpatients with community-acquired pneumonia; 2) pediatric inpatients with community-acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media.

DETAILED DESCRIPTION:
Antibiotic stewardship has been shown to improve patient outcomes, decrease adverse events, and decrease antibiotic resistance. This group of investigators previously partnered with collaborators at the Centers for Disease Control and Prevention and conducted relevant pilot work in developing and validating electronic indicators of inappropriate antibiotic prescribing for 8 conditions, amongst which are the four conditions of interest in this study: adult inpatients with community-acquired pneumonia; pediatric inpatients with community-acquired pneumonia; adult outpatients with acute pharyngitis; and pediatric outpatients with acute otitis media. Methods were developed to generate automatic, routine reports to identify elements of inappropriate antibiotic use including; 1) the decision to initiate antibiotic therapy (pharyngitis and acute otitis media only); 2) the choice of antibiotic agent; and 3) the duration of antibiotic use.

The purpose of this project is to assess the impact of these developed electronic indicators on supporting antibiotic stewardship efforts to improve the appropriateness of antibiotic use, as well as the acceptability and feasibility of delivering these reports to prescribers. The investigators aim to:

1. Refine and validate indicators of appropriate antibiotic use by utilizing Electronic Health Record data, including International Classification of Diseases version 10 codes, medications, laboratory data, co-morbid medical conditions, site of care, clinical documentation, prior hospitalizations, and medication exposure. The researchers will validate the definitions of the various conditions and appropriateness captured electronically with a manual chart review of clinical documentation.
2. Implement a scalable and sustainable antimicrobial stewardship feedback report-based intervention for these four conditions informed by a rapid user-centered design process.
3. Track the impact of the stewardship interventions and report to key stakeholders, including prescribers.
4. Create a publicly available toolkit based on the findings of this project that includes: (i) analytic tools and resources for using the automated reports of key indicators to target stewardship interventions and (ii) an implementation guide to inform the application of automated reports to stewardship in the inpatient and outpatient settings.

If proven effective, these electronic health record-based approaches hold the promise to greatly enhance the effectiveness and efficiency of antimicrobial stewardship initiatives.

ELIGIBILITY:
Patient Inclusion Criteria:

* Diagnosis of one of four conditions based on ICD-10 diagnostic codes.

Patient Exclusion Criteria:

* Presence of specific complex chronic conditions
* Use of immunocompromising medications
* Transfer from another health facility.

Clinician Inclusion Criteria:

* Prescribing clinicians (including attending physicians, fellows, residents, nurse practitioners, and physician assistants) at one of the participating outpatient practices or inpatient units.
* Age ≥ 18 years old
* Employed by one of the participating sites

Clinician Exclusion Criteria:

* Volunteers or other non-employee hospital staff
* Limited English proficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26139 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
This study was initiated prior to the NIH Data Management and Sharing Policy update that was released on January 25, 2023.

REFERENCES:
- [Background] Gerber JS, Newland JG, Coffin SE, Hall M, Thurm C, Prasad PA, Feudtner C, Zaoutis TE. Variability in antibiotic use at children's hospitals. Pediatrics. 2010 Dec;126(6):1067-73. doi: 10.1542/peds.2010-1275. Epub 2010 Nov 15. PMID 21078728
- [Background] Polk RE, Hohmann SF, Medvedev S, Ibrahim O. Benchmarking risk-adjusted adult antibacterial drug use in 70 US academic medical center hospitals. Clin Infect Dis. 2011 Dec;53(11):1100-10. doi: 10.1093/cid/cir672. Epub 2011 Oct 13. PMID 21998281
- [Background] Roberts RM, Hicks LA, Bartoces M. Variation in US outpatient antibiotic prescribing quality measures according to health plan and geography. Am J Manag Care. 2016 Aug;22(8):519-23. PMID 27541698
- [Background] Hicks LA, Bartoces MG, Roberts RM, Suda KJ, Hunkler RJ, Taylor TH Jr, Schrag SJ. US outpatient antibiotic prescribing variation according to geography, patient population, and provider specialty in 2011. Clin Infect Dis. 2015 May 1;60(9):1308-16. doi: 10.1093/cid/civ076. Epub 2015 Mar 5. PMID 25747410
- [Background] Barnett ML, Linder JA. Antibiotic prescribing for adults with acute bronchitis in the United States, 1996-2010. JAMA. 2014 May 21;311(19):2020-2. doi: 10.1001/jama.2013.286141. No abstract available. PMID 24846041
- [Background] Barnett ML, Linder JA. Antibiotic prescribing to adults with sore throat in the United States, 1997-2010. JAMA Intern Med. 2014 Jan;174(1):138-40. doi: 10.1001/jamainternmed.2013.11673. No abstract available. PMID 24091806
- [Background] Fairlie T, Shapiro DJ, Hersh AL, Hicks LA. National trends in visit rates and antibiotic prescribing for adults with acute sinusitis. Arch Intern Med. 2012 Oct 22;172(19):1513-4. doi: 10.1001/archinternmed.2012.4089. No abstract available. PMID 23007315
- [Background] Fleming-Dutra KE, Hersh AL, Shapiro DJ, Bartoces M, Enns EA, File TM Jr, Finkelstein JA, Gerber JS, Hyun DY, Linder JA, Lynfield R, Margolis DJ, May LS, Merenstein D, Metlay JP, Newland JG, Piccirillo JF, Roberts RM, Sanchez GV, Suda KJ, Thomas A, Woo TM, Zetts RM, Hicks LA. Prevalence of Inappropriate Antibiotic Prescriptions Among US Ambulatory Care Visits, 2010-2011. JAMA. 2016 May 3;315(17):1864-73. doi: 10.1001/jama.2016.4151. PMID 27139059
- [Background] Dellit TH, Owens RC, McGowan JE Jr, Gerding DN, Weinstein RA, Burke JP, Huskins WC, Paterson DL, Fishman NO, Carpenter CF, Brennan PJ, Billeter M, Hooton TM; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. Clin Infect Dis. 2007 Jan 15;44(2):159-77. doi: 10.1086/510393. Epub 2006 Dec 13. No abstract available. PMID 17173212
- [Background] Gerber JS, Grundmeier R, Hamilton KW, Hicks L, Neuhauser M, Frager N, Menon M, Kratz E, Jaskowiak A, Cressman L, James T, Omorogbe J, Lautenbach E. Development of an Electronic Algorithm to Identify Inappropriate Antibiotic Prescribing for Pediatric Pharyngitis. Infection Control and Hospital Epidemiology. 2020;41 (S1):S188-189
- [Background] Gerber JS, Grundmeier R, Hamilton KW, Hicks L, Neuhauser M, Frager N, Menon M, Kratz E, Jaskowiak A, Cressman L, James T, Omorogbe J, Lautenbach E. An Electronic Algorithm to Better Target Antimicrobial Stewardship Program (ASP) Efforts for Children Hospitalized with Community-Acquired Pneumonia (CAP). Open Forum Infectious Diseases. 2020;7 (S1):S85-86
- [Background] Lautenbach E, Hamilton KH, Grundmeier R, Neuhauser M, Hicks L, Jaskowiak A, Cressman L, James T, Omorogbe J, Frager N, Menon M, Kratz E, Gerber JS. Development of an Electronic Algorithm to Target Outpatient Antimicrobial Stewardship Efforts for Acute Bronchitis. Infection Control and Hospital Epidemiology. 2020;41 (S1):S188-189
- [Background] Lautenbach E, Hamilton KW, Grundmeier R, Neuhauser MM, Hicks LA, Jaskowiak-Barr A, Cressman L, James T, Omorogbe J, Frager N, Menon M, Kratz E, Dutcher L, Chiotos K, Gerber JS. Development of an Electronic Algorithm to Target Outpatient Antimicrobial Stewardship Efforts for Acute Bronchitis and Pharyngitis. Open Forum Infect Dis. 2022 Jun 6;9(7):ofac273. doi: 10.1093/ofid/ofac273. eCollection 2022 Jul. PMID 35854991
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Background] Charani E, Ahmad R, Rawson TM, Castro-Sanchez E, Tarrant C, Holmes AH. The Differences in Antibiotic Decision-making Between Acute Surgical and Acute Medical Teams: An Ethnographic Study of Culture and Team Dynamics. Clin Infect Dis. 2019 Jun 18;69(1):12-20. doi: 10.1093/cid/ciy844. PMID 30445453
- [Background] Szymczak JE. Are Surgeons Different? The Case for Bespoke Antimicrobial Stewardship. Clin Infect Dis. 2019 Jun 18;69(1):21-23. doi: 10.1093/cid/ciy847. No abstract available. PMID 30445615
- [Background] Landis-Lewis Z, Kononowech J, Scott WJ, Hogikyan RV, Carpenter JG, Periyakoil VS, Miller SC, Levy C, Ersek M, Sales A. Designing clinical practice feedback reports: three steps illustrated in Veterans Health Affairs long-term care facilities and programs. Implement Sci. 2020 Jan 21;15(1):7. doi: 10.1186/s13012-019-0950-y. PMID 31964414
- [Background] Redding LE, Muller BM, Szymczak JE. Small and Large Animal Veterinarian Perceptions of Antimicrobial Use Metrics for Hospital-Based Stewardship in the United States. Front Vet Sci. 2020 Sep 8;7:582. doi: 10.3389/fvets.2020.00582. eCollection 2020. PMID 33102546
- [Background] Szymczak JE, Feemster KA, Zaoutis TE, Gerber JS. Pediatrician perceptions of an outpatient antimicrobial stewardship intervention. Infect Control Hosp Epidemiol. 2014 Oct;35 Suppl 3:S69-78. doi: 10.1086/677826. PMID 25222901
- [Background] Szymczak JE, Kitt E, Hayes M, Chiotos K, Coffin SE, Schriver ER, Patton AM, Metjian TA, Gerber JS. Threatened efficiency not autonomy: Prescriber perceptions of an established pediatric antimicrobial stewardship program. Infect Control Hosp Epidemiol. 2019 May;40(5):522-527. doi: 10.1017/ice.2019.47. Epub 2019 Mar 28. PMID 30919799
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Result] Chiotos K, Dutcher L, Grundmeier RW, Meyahnwi D, Lautenbach E, Neuhauser MM, Hicks LA, Hamilton KW, Li Y, Szymczak JE, Muller BM, Congdon M, Kane E, Hart J, Utidjian L, Cressman L, Jaskowiak-Barr A, Gerber JS. Impact of Clinician Feedback Reports on Antibiotic Use in Children Hospitalized With Community-acquired Pneumonia. Clin Infect Dis. 2025 Feb 24;80(2):263-270. doi: 10.1093/cid/ciae593. PMID 39656188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with one or more of the target conditions during the study period were included.
Pre-assignment Details: Clinicians were not enrolled as participants diagnosed with conditions of interest during the pre-intervention and post-intervention study periods. The clinicians were administered a survey once during the post-intervention period.
Groups:
- Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period: This study evaluates changes in antibiotic prescribing practices following a stewardship intervention. The pre intervention time period defines the baseline cohort of patients diagnosed with one of the four target conditions, before exposure to the stewardship intervention.
- Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period: This study evaluates changes in antibiotic prescribing practices following a stewardship intervention. The post-intervention time period defines the cohort of patients diagnosed with one of the four target conditions, after exposure to the stewardship intervention.
Period: Overall Study
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Started | 12917 | 13222
Adult Inpatients With Community Acquired Pneumonia | 305 | 330
Pediatric Inpatients With Community Acquired Pneumonia | 413 | 387
Adult Outpatients With Pharyngitis | 2032 | 3764
Pediatric Outpatients With Acute Otitis Media (Outcome measures for overall guideline-concordant antibiotic use, guideline-concordant antibiotic choice, and guideline-concordant antibiotic duration are measured only in subset of participants who were prescribed antibiotics - 9,020 participants in pre-intervention period and 7,778 participants in the post-intervention period.) | 10167 | 8741
Completed | 12917 | 13222
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Total
Number analyzed (Participants) | 12917 | 13222 | 26139
Age, Categorical [Count of Participants; unit: Participants] — Population: The pre-intervention and post-intervention cohort of patients are diagnosed with one of the four target conditions. The four population sub-groups are 1) adult inpatients with community acquired pneumonia; 2) pediatric inpatients with community acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media, which are noted with different row populations based on condition.
  Participants
    Total: <=18 years | 10628 | 9177 | 19805
    Total: Between 18 and 65 years | 1838 | 3341 | 5179
    Total: >=65 years | 451 | 704 | 1155
    Adult Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 305 | 330 | 635
    Adult Inpatients With Community Acquired Pneumonia: <=18 years | 0 | 0 | 0
    Adult Inpatients With Community Acquired Pneumonia: Between 18 and 65 years | 173 | 182 | 355
    Adult Inpatients With Community Acquired Pneumonia: >=65 years | 132 | 148 | 280
    Pediatric Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 413 | 387 | 800
    Pediatric Inpatients With Community Acquired Pneumonia: <=18 years | 413 | 387 | 800
    Pediatric Inpatients With Community Acquired Pneumonia: Between 18 and 65 years | 0 | 0 | 0
    Pediatric Inpatients With Community Acquired Pneumonia: >=65 years | 0 | 0 | 0
    Adult Outpatients With Pharyngitis: number analyzed (Participants) | 2032 | 3764 | 5796
    Adult Outpatients With Pharyngitis: <=18 years | 48 | 49 | 97
    Adult Outpatients With Pharyngitis: Between 18 and 65 years | 1665 | 3159 | 4824
    Adult Outpatients With Pharyngitis: >=65 years | 319 | 556 | 875
    Pediatric Outpatients With Acute Otitis Media: number analyzed (Participants) | 10167 | 8741 | 18908
    Pediatric Outpatients With Acute Otitis Media: <=18 years | 10167 | 8741 | 18908
    Pediatric Outpatients With Acute Otitis Media: Between 18 and 65 years | 0 | 0 | 0
    Pediatric Outpatients With Acute Otitis Media: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The pre-intervention and post-intervention cohort of patients are diagnosed with one of the four target conditions. The four population sub-groups are 1) adult inpatients with community acquired pneumonia; 2) pediatric inpatients with community acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media, which are noted with different row populations based on condition.
  Participants
    Total: Female | 6522 | 7215 | 13737
    Total: Male | 6395 | 6007 | 12402
    Adult Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 305 | 330 | 635
    Adult Inpatients With Community Acquired Pneumonia: Female | 168 | 178 | 346
    Adult Inpatients With Community Acquired Pneumonia: Male | 137 | 152 | 289
    Pediatric Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 413 | 387 | 800
    Pediatric Inpatients With Community Acquired Pneumonia: Female | 204 | 195 | 399
    Pediatric Inpatients With Community Acquired Pneumonia: Male | 209 | 192 | 401
    Adult Outpatients With Pharyngitis: number analyzed (Participants) | 2032 | 3764 | 5796
    Adult Outpatients With Pharyngitis: Female | 1436 | 2709 | 4145
    Adult Outpatients With Pharyngitis: Male | 596 | 1055 | 1651
    Pediatric Outpatients With Acute Otitis Media: number analyzed (Participants) | 10167 | 8741 | 18908
    Pediatric Outpatients With Acute Otitis Media: Female | 4714 | 4132 | 8846
    Pediatric Outpatients With Acute Otitis Media: Male | 5453 | 4609 | 10062
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The pre-intervention and post-intervention cohort of patients are diagnosed with one of the four target conditions. The four population sub-groups are 1) adult inpatients with community acquired pneumonia; 2) pediatric inpatients with community acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media, which are noted with different row populations based on condition.
  Participants
    Total: Hispanic or Latino | 889 | 924 | 1813
    Total: Not Hispanic or Latino | 11885 | 12020 | 23905
    Total: Unknown or Not Reported | 143 | 278 | 421
    Adult Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 305 | 330 | 635
    Adult Inpatients With Community Acquired Pneumonia: Hispanic or Latino | 9 | 9 | 18
    Adult Inpatients With Community Acquired Pneumonia: Not Hispanic or Latino | 296 | 320 | 616
    Adult Inpatients With Community Acquired Pneumonia: Unknown or Not Reported | 0 | 1 | 1
    Pediatric Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 413 | 387 | 800
    Pediatric Inpatients With Community Acquired Pneumonia: Hispanic or Latino | 69 | 59 | 128
    Pediatric Inpatients With Community Acquired Pneumonia: Not Hispanic or Latino | 339 | 317 | 656
    Pediatric Inpatients With Community Acquired Pneumonia: Unknown or Not Reported | 5 | 11 | 16
    Adult Outpatients With Pharyngitis: number analyzed (Participants) | 2032 | 3764 | 5796
    Adult Outpatients With Pharyngitis: Hispanic or Latino | 101 | 185 | 286
    Adult Outpatients With Pharyngitis: Not Hispanic or Latino | 1911 | 3529 | 5440
    Adult Outpatients With Pharyngitis: Unknown or Not Reported | 20 | 50 | 70
    Pediatric Outpatients With Acute Otitis Media: number analyzed (Participants) | 10167 | 8741 | 18908
    Pediatric Outpatients With Acute Otitis Media: Hispanic or Latino | 710 | 671 | 1381
    Pediatric Outpatients With Acute Otitis Media: Not Hispanic or Latino | 9339 | 7854 | 17193
    Pediatric Outpatients With Acute Otitis Media: Unknown or Not Reported | 118 | 216 | 334
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The pre-intervention and post-intervention cohort of patients are diagnosed with one of the four target conditions. The four population sub-groups are 1) adult inpatients with community acquired pneumonia; 2) pediatric inpatients with community acquired pneumonia; 3) adult outpatients with acute pharyngitis; and 4) pediatric outpatients with acute otitis media, which are noted with different row populations based on condition.
  Participants
    Total: American Indian or Alaska Native | 5 | 6 | 11
    Total: Asian | 306 | 393 | 699
    Total: Native Hawaiian or Other Pacific Islander | 7 | 12 | 19
    Total: Black or African American | 1701 | 1825 | 3526
    Total: White | 9110 | 9058 | 18168
    Total: More than one race | 360 | 391 | 751
    Total: Unknown or Not Reported | 1428 | 1537 | 2965
    Adult Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 305 | 330 | 635
    Adult Inpatients With Community Acquired Pneumonia: American Indian or Alaska Native | 0 | 2 | 2
    Adult Inpatients With Community Acquired Pneumonia: Asian | 6 | 8 | 14
    Adult Inpatients With Community Acquired Pneumonia: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adult Inpatients With Community Acquired Pneumonia: Black or African American | 203 | 209 | 412
    Adult Inpatients With Community Acquired Pneumonia: White | 81 | 89 | 170
    Adult Inpatients With Community Acquired Pneumonia: More than one race | 3 | 2 | 5
    Adult Inpatients With Community Acquired Pneumonia: Unknown or Not Reported | 12 | 20 | 32
    Pediatric Inpatients With Community Acquired Pneumonia: number analyzed (Participants) | 413 | 387 | 800
    Pediatric Inpatients With Community Acquired Pneumonia: American Indian or Alaska Native | 0 | 0 | 0
    Pediatric Inpatients With Community Acquired Pneumonia: Asian | 21 | 23 | 44
    Pediatric Inpatients With Community Acquired Pneumonia: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Pediatric Inpatients With Community Acquired Pneumonia: Black or African American | 130 | 117 | 247
    Pediatric Inpatients With Community Acquired Pneumonia: White | 171 | 158 | 329
    Pediatric Inpatients With Community Acquired Pneumonia: More than one race | 19 | 19 | 38
    Pediatric Inpatients With Community Acquired Pneumonia: Unknown or Not Reported | 71 | 70 | 141
    Adult Outpatients With Pharyngitis: number analyzed (Participants) | 2032 | 3764 | 5796
    Adult Outpatients With Pharyngitis: American Indian or Alaska Native | 1 | 4 | 5
    Adult Outpatients With Pharyngitis: Asian | 74 | 152 | 226
    Adult Outpatients With Pharyngitis: Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
    Adult Outpatients With Pharyngitis: Black or African American | 312 | 550 | 862
    Adult Outpatients With Pharyngitis: White | 1477 | 2724 | 4201
    Adult Outpatients With Pharyngitis: More than one race | 24 | 40 | 64
    Adult Outpatients With Pharyngitis: Unknown or Not Reported | 141 | 290 | 431
    Pediatric Outpatients With Acute Otitis Media: number analyzed (Participants) | 10167 | 8741 | 18908
    Pediatric Outpatients With Acute Otitis Media: American Indian or Alaska Native | 4 | 0 | 4
    Pediatric Outpatients With Acute Otitis Media: Asian | 205 | 210 | 415
    Pediatric Outpatients With Acute Otitis Media: Native Hawaiian or Other Pacific Islander | 3 | 8 | 11
    Pediatric Outpatients With Acute Otitis Media: Black or African American | 1056 | 949 | 2005
    Pediatric Outpatients With Acute Otitis Media: White | 7381 | 6087 | 13468
    Pediatric Outpatients With Acute Otitis Media: More than one race | 314 | 330 | 644
    Pediatric Outpatients With Acute Otitis Media: Unknown or Not Reported | 1204 | 1157 | 2361

OUTCOME MEASURES:

1. Primary Outcome: Guideline-concordant Antibiotic Use for Adults With Pharyngitis
Description: Count of participants with pharyngitis with guideline-concordant antibiotic use for all three metrics (decision to prescribe an antibiotic, antibiotic choice, and antibiotic duration). The count of participants with pharyngitis with guideline-concordant antibiotic use for all three metrics was divided by the total number of participants with pharyngitis to generate the percentage of participants receiving guideline-concordant antibiotic use for all three metrics. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for adults with pharyngitis only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 2032 | 3764
Participants | 1458 | 2477

2. Primary Outcome: Guideline-concordant Antibiotic Use for Children With Acute Otitis Media
Description: Count of participants with acute otitis media with guideline-concordant antibiotic use for all three metrics (decision to prescribe an antibiotic, antibiotic choice, and antibiotic duration). The count of participants with acute otitis media with guideline-concordant antibiotic use for all three metrics was divided by the total number of participants with pediatric acute otitis media who were prescribed antibiotics to generate the percentage of participants receiving guideline-concordant antibiotic use for all three metrics. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Note: this metric of guideline-concordant antibiotic use was measured using a denominator of those who were prescribed antibiotics (pre-intervention: 9,020 participants; post-intervention: 7,778 participants). The overall number of participants with acute otitis media (pre-intervention: 10,167 participants; post-intervention: 8,741 participants) was NOT used as the denominator for this reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 9020 | 7778
Participants | 6154 | 6287

3. Primary Outcome: Guideline-concordant Antibiotic Use for Adults With Community-acquired Pneumonia
Description: Count of participants with community-acquired pneumonia with guideline-concordant antibiotic use for all three metrics (decision to prescribe an antibiotic, antibiotic choice, and antibiotic duration). The count of participants with community-acquired pneumonia with guideline-concordant antibiotic use for all three metrics was divided by the total number of participants with community-acquired pneumonia to generate the percentage of participants receiving guideline-concordant antibiotic use for all three metrics. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for adults with community-acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 305 | 330
Participants | 204 | 242

4. Primary Outcome: Guideline-concordant Antibiotic Use for Children With Community-acquired Pneumonia
Description: Count of participants with pediatric community-acquired pneumonia with guideline-concordant antibiotic use for all three metrics (decision to prescribe an antibiotic, antibiotic choice, and antibiotic duration). The count of participants with pediatric community-acquired pneumonia with guideline-concordant antibiotic use for all three metrics was divided by the total number of participants with pediatric community-acquired pneumonia to generate the percentage of participants receiving guideline-concordant antibiotic use for all three metrics. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for children with community-acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 413 | 387
Participants | 213 | 308

5. Secondary Outcome: Guideline-concordant Antibiotic Choice for Adults Hospitalized With Community Acquired Pneumonia
Description: Count of participants with community-acquired pneumonia with guideline-concordant antibiotic use for antibiotic choice. The count of participants with community-acquired pneumonia with guideline-concordant antibiotic use for this metric was divided by the total number of participants with community-acquired pneumonia to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic choice. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for adults hospitalized with community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 305 | 330
Participants | 268 | 302

6. Secondary Outcome: Guideline-concordant Antibiotic Duration for Adults Hospitalized With Community Acquired Pneumonia
Description: Count of participants with community-acquired pneumonia with guideline-concordant antibiotic use for antibiotic duration. The count of participants with community-acquired pneumonia with guideline-concordant antibiotic use for this metric was divided by the total number of participants with community-acquired pneumonia to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic duration. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for adults hospitalized with community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 305 | 330
Participants | 230 | 261

7. Secondary Outcome: 30-day Community Acquired Pneumonia-related Outpatient Revisits (Emergency Department, Urgent Care, or Primary Care) in Adults
Description: Count of participants with community-acquired pneumonia with a return visit in the outpatient setting (emergency department, urgent care, or primary care) for community acquired pneumonia within 30 days of discharge following index hospitalization for adult community acquired pneumonia. The count of participants with community-acquired pneumonia with a return visit in the outpatient setting was divided by the total number of participants with community-acquired pneumonia to generate the percentage of participants with a return visit in the outpatient setting.
Time Frame: 30 days
Population: Data for adults with community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 305 | 330
Participants | 0 | 0

8. Secondary Outcome: 30-day Readmissions for Community Acquired Pneumonia in Adults
Description: Count of participants with a readmission for community-acquired pneumonia within 30 days of discharge following an index hospitalization for community-acquired pneumonia. The count of participants with a readmission for community-acquired pneumonia was divided by the total number of participants with community-acquired pneumonia to generate the percentage of participants with readmissions within 30 days of discharge following an index hospitalization for community-acquired pneumonia.
Time Frame: 30 days
Population: Data for adults with community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 305 | 330
Participants | 13 | 6

9. Secondary Outcome: Guideline-concordant Antibiotic Choice for Pediatric Community Acquired Pneumonia
Description: Count of participants with pediatric community-acquired pneumonia with guideline-concordant antibiotic use for antibiotic choice. The count of participants with pediatric community-acquired pneumonia with guideline-concordant antibiotic use for this metric was divided by the total number of participants with pediatric community-acquired pneumonia to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic choice. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for pediatric community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 413 | 387
Participants | 394 | 362

10. Secondary Outcome: Guideline-concordant Antibiotic Duration for Pediatric Community Acquired Pneumonia
Description: Count of participants with pediatric community-acquired pneumonia with guideline-concordant antibiotic use for antibiotic duration. The count of participants with pediatric community-acquired pneumonia with guideline-concordant antibiotic use for this metric was divided by the total number of participants with pediatric community-acquired pneumonia to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic duration. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for pediatric community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 413 | 387
Participants | 221 | 322

11. Secondary Outcome: 28-day Community Acquired Pneumonia-related Outpatient Revisits (Emergency Department, Urgent Care, or Primary Care) in Children
Description: Count of participants with pediatric community-acquired pneumonia with a return visit in the outpatient setting (emergency department, urgent care, or primary care) for pediatric community acquired pneumonia within 28 days of discharge following index hospitalization for pediatric community acquired pneumonia. The count of participants with pediatric community-acquired pneumonia with a return visit in the outpatient setting was divided by the total number of participants with pediatric community-acquired pneumonia to generate the percentage of participants with a return visit in the outpatient setting.
Time Frame: 28 days
Population: Data for pediatric community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 413 | 387
Participants | 13 | 20

12. Secondary Outcome: 28-day Readmissions for Pediatric Community Acquired Pneumonia
Description: Count of participants with a readmission for community-acquired pneumonia within 28 days of discharge following an index hospitalization for community-acquired pneumonia. The count of participants with a readmission for community-acquired pneumonia was divided by the total number of participants with community-acquired pneumonia to generate the percentage of participants with readmissions within 28 days of discharge following an index hospitalization for community-acquired pneumonia.
Time Frame: 28 days
Population: Data for pediatric community acquired pneumonia only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 413 | 387
Participants | 8 | 14

13. Secondary Outcome: Guideline-concordant Decision to Prescribe Antibiotics for Adult Pharyngitis
Description: Count of participants with pharyngitis for which the decision to prescribe an antibiotic was correct. The count of participants with pharyngitis for which the decision to prescribe an antibiotic was correct was divided by the total number of participants with pharyngitis to generate the percentage of participants for which the decision to prescribe an antibiotic was correct. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: This metric encapsulates patients who did and did not receive antibiotics.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 2032 | 3764
Participants | 1464 | 2492

14. Secondary Outcome: Guideline-concordant Antibiotic Choice Adult Pharyngitis
Description: Count of participants with adult pharyngitis with guideline-concordant antibiotic use for antibiotic choice. The count of participants with pharyngitis with guideline-concordant antibiotic use for this metric was divided by the total number of participants with pharyngitis to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic choice. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Note: this metric of guideline-concordant antibiotic use was measured using a denominator of those who were prescribed antibiotics for adult pharyngitis (pre-intervention: 32 participants; post-intervention: 175 participants). The overall number of participants with adult pharyngitis (pre-intervention: 2,032 participants; post-intervention: 3,764 participants) was NOT used as the denominator for this reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 32 | 175
Participants | 27 | 160

15. Secondary Outcome: Guideline-concordant Antibiotic Duration for Adult Pharyngitis
Description: Count of participants with adult pharyngitis with guideline-concordant antibiotic use for antibiotic duration. The count of participants with pharyngitis with guideline-concordant antibiotic use for this metric was divided by the total number of participants with pharyngitis to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic duration. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 32 | 175
Participants | 31 | 175

16. Secondary Outcome: 30-day Pharyngitis Outpatient Revisits (Emergency Department, Urgent Care, or Primary Care) in Adults
Description: Count of participants with adult pharyngitis with a return visit in the outpatient setting (emergency department, urgent care, or primary care) for pharyngitis within 30 days of discharge following index hospitalization for adult pharyngitis. The count of participants with pharyngitis with a return visit in the outpatient setting was divided by the total number of participants with pharyngitis to generate the percentage of participants with a return visit in the outpatient setting.
Time Frame: 30 days
Population: Data for Adult Pharyngitis only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 2032 | 3764
Participants | 291 | 578

17. Secondary Outcome: 30-day Deep Neck Space Infection Admission
Description: Count of participants with a readmission for deep neck space infection within 30 days of index encounter for pharyngitis. The count of participants with a readmission for deep neck space infection was divided by the total number of participants with adult pharyngitis to generate the percentage of participants with readmissions for deep neck space infection within 30 days of index encounter for pharyngitis.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 2032 | 3764
Participants | 0 | 1

18. Secondary Outcome: Guideline-concordant Decision to Prescribe Antibiotics for Pediatric Acute Otitis Media
Description: Count of participants with pediatric acute otitis media for which the decision to prescribe an antibiotic was correct. The count of participants with pediatric acute otitis media for which the decision to prescribe an antibiotic was correct was divided by the total number of participants with pediatric acute otitis media to generate the percentage of participants for which the decision to prescribe an antibiotic was correct. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: This metric encapsulates patients who did and did not receive antibiotics.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 10167 | 8741
Participants | 9935 | 8547

19. Secondary Outcome: Guideline-concordant Antibiotic Choice for Pediatric Acute Otitis Media
Description: Count of participants with pediatric acute otitis media with guideline-concordant antibiotic use for antibiotic choice. The count of participants with pediatric acute otitis media visits with guideline-concordant antibiotic use for this metric was divided by the total number of participants with pediatric acute otitis media who were prescribed antibiotics to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic choice. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for pediatric acute otitis media only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 9020 | 7778
Participants | 7498 | 6828

20. Secondary Outcome: Guideline-concordant Antibiotic Duration for Pediatric Acute Otitis Media
Description: Count of participants with pediatric acute otitis media with guideline-concordant antibiotic use for antibiotic duration. The count of participants with pediatric acute otitis media with guideline-concordant antibiotic use for this metric was divided by the total number of participants with pediatric acute otitis media who were prescribed antibiotics to generate the percentage of participants receiving guideline-concordant antibiotic use for antibiotic duration. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Data for pediatric acute otitis media only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 9020 | 7778
Participants | 7565 | 7281

21. Secondary Outcome: 28-day Acute Otitis Media-related Outpatient Revisits (Emergency Department, Urgent Care, or Primary Care)
Description: Count of participants with pediatric acute otitis media with a return visit in the outpatient setting (emergency department, urgent care, or primary care) for pediatric acute otitis media within 28 days of the index acute otitis media encounter. The count of participants with pediatric acute otitis media with a return visit in the outpatient setting was divided by the total number of participants with pediatric acute otitis media to generate the percentage of participants with a return visit in the outpatient setting.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 10167 | 8741
Participants | 891 | 756

22. Secondary Outcome: 28-day Mastoiditis or Intracranial Infection Admissions
Description: Count of participants with a readmission for mastoiditis or intracranial infection within 28 days of the index encounter for pediatric acute otitis media. The count of participants with a readmission for mastoiditis or intracranial infection was divided by the total number of participants with pediatric acute otitis media to generate the percentage of participants with readmissions within 28 days of discharge following an index hospitalization for acute otitis media.
Time Frame: 28 days
Population: Data for pediatric acute otitis media only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 10167 | 8741
Participants | 0 | 0

23. Secondary Outcome: Guideline-concordant Decision to Not Prescribe Antibiotics for Pediatric Acute Otitis Media
Description: Count of participants with pediatric acute otitis media with guideline-concordant antibiotic use for appropriate decision not to prescribe antibiotics. The count of participants with pediatric acute otitis media with an appropriate decision not to prescribe antibiotics was divided by the total number of participants with no antibiotics prescribed to generate the percentage of participants appropriately not prescribed antibiotics for acute otitis media. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Of note, only a subgroup of patients were assessed with this metric.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 1155 | 983
Participants | 284 | 292

24. Secondary Outcome: Guideline-concordant Decision to Not Prescribe Antibiotics for Adult Pharyngitis
Description: Count of participants with adult pharyngitis with guideline-concordant antibiotic use for appropriate decision not to prescribe antibiotics. The count of participants with adult pharyngitis with an appropriate decision not to prescribe antibiotics was divided by the total number of participants with no antibiotics prescribed to generate the percentage of participants appropriately not prescribed antibiotics for pharyngitis. These proportions were compared for the group of participants in the pre intervention period (1 year) and the post intervention period (1 year). There were not individual participant level measures for this outcome.
Time Frame: Pre-intervention and post-intervention, up to 2 years
Population: Of note, only a subgroup of patients were assessed with this metric.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
Number analyzed (Participants) | 1432 | 2317
Participants | 1432 | 2312

25. Other Pre Specified Outcome: Feasibility of Intervention - Outpatient
Description: Feasibility is defined as the extent to which the intervention can be carried out in the clinical setting. The feasibility of intervention measure is the full name of this scale. The feasibility of intervention scale consists of four questions, each with 5 possible responses (completely disagree, disagree, neither agree or disagree, agree, or completely agree) on a numeric 1-5 scale. These four subscores are summed to generate a total score, with possible scores ranging from 4-20. A higher score indicates that the intervention is more feasible. There are no validated cutoffs for feasibility. The mean total score and standard deviation of the mean total score for all respondents are reported. The feasibility of intervention measure was assessed by a one time survey in the post-intervention time period.
Time Frame: One time measure in the post intervention time period
Population: The pre-intervention and post-intervention clinicians are the same people and this survey was administered to this group of individuals once during the post-intervention period.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Outpatient Clinicians: We surveyed clinicians receiving the pharyngitis and acute otitis media reports to understand feasibility and acceptability.
Arm/Group | Outpatient Clinicians
Number analyzed (Participants) | 45
units on a scale | 15.7 (3.1)

26. Other Pre Specified Outcome: Acceptability of Intervention - Outpatient
Description: Acceptability is defined as how well the intervention was received by the prescribing clinicians. The acceptability of intervention measure is the full name of this scale. The acceptability of intervention scale consists of four questions, each with 5 possible responses (completely disagree, disagree, neither agree or disagree, agree, or completely agree) on a numeric 1-5 scale. These four subscores are summed to generate a total score, with possible scores ranging from 4-20. A higher score indicates that the intervention is more acceptable. There are no validated cutoffs for acceptability. The mean total score and standard deviation of the mean total score for all respondents are reported. The acceptability of intervention measure was assessed by a one time survey in the post-intervention time period.
Time Frame: One time measure in the post intervention time period
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outpatient Clinicians
Number analyzed (Participants) | 45
units on a scale | 13.4 (4.6)

27. Other Pre Specified Outcome: Feasibility of Intervention Measure - Inpatient
Description: as for outcome 25
Time Frame: One time measure in the post intervention time period
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Postintervention: $
Arm/Group | Preintervention | Postintervention
Number analyzed (Participants) | 0 | 36
units on a scale |  | 17.7 (3.1)

28. Other Pre Specified Outcome: Acceptability of Intervention Measure - Inpatient
Description: as for outcome 26
Time Frame: One time measure in the post intervention time period.
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inpatient Clinicians: We surveyed inpatient clinicians receiving the community acquired pneumonia reports to understand feasibility and acceptability of the measures.
Arm/Group | Inpatient Clinicians
Number analyzed (Participants) | 36
units on a scale | 17.2 (3.5)

ADVERSE EVENTS:
Time Frame: This was a minimal risk study deemed exempt research by the CHOP and UPenn IRB. Serious adverse events, non-serious adverse events, and mortality were not collected in this study.
Description: This was a minimal risk study deemed exempt research by the CHOP and UPenn IRB. Serious adverse events, non-serious adverse events, and mortality were not collected in this study.
Arm/Group | Pre-Intervention: Patients Diagnosed With Conditions of Interest During Study Period | Post-Intervention: Patients Diagnosed With Conditions of Interest During Study Period
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT06027593/Prot_SAP_000.pdf